CLINICAL TRIAL: NCT03218540
Title: Directed Fluid Therapy Based on Stroke Volume Variations Improves Fluid Management in Endovascular Aortic Repair for Aortic Aneurysm Patients: a Randomized Trial
Brief Title: Stroke Volume Variation vs Central Venous Pressure Guidance Fluid Management in Endovascular Aortic Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE591258
Record Dates: First submitted 2017-07-10; First posted 2017-07-14 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Complications
Keywords: stroke volume variation; central venous pressure; serum lactate; serum creatinine
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Group SVV: fluid management guided by stroke volume variation (SVV) protocol Group CVP: fluid management guided by central venous pressure (CVP) protocol
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient is anesthetized, thus unaware type of treatment. The assessor is blinded of the monitor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SVV group (Experimental): Fluid management protocol
  Interventions: Procedure: Fluid management protocol
- CVP group (Active Comparator): Fluid management protocol
  Interventions: Procedure: Fluid management protocol

INTERVENTIONS:
Procedure: Fluid management protocol — SVV protocol: keep SVV 10-13% and give fluid when SVV > 13% CVP protocol: keep CVP 8-12 mmHG and give fluid when CVP < 8 mmHg

SUMMARY:
Hypothesis: Fluid management guided by stroke volume variation (SVV), compared with central venous pressure (CVP), guidance results in better clinical outcomes.

Primary outcomes: Perioperative, up to 48 h postoperative, serum lactate and creatinine level.

Methods: Adult patients undergoing endovascular aortic aneurysm repair (EVAR) will be randomized into 2 groups: SVV group managed by SVV guidance and CVP group managed by CVP guidance.

Outcome analyses: Compare serum lactate, creatinine as well as other postoperative complications between both groups.

DETAILED DESCRIPTION:
Objective: To compare postoperative clinical outcome in adult patient undergoing EVAR.

Primary outcome: Postoperative serum lactate and creatinine.

Secondary outcome: Postoperative complications.

Methods: Eligible patients will be randomized to 2 groups. Both groups will be managed intraoperatively in the same way, except fluid management protocol. SVV group will be managed according to stroke volume variation (SVV) protocol, i.e., control SVV 10-13% and give fluid when SVV > 13%. CVP group will be managed using central venous pressure (CVP) protocol, i.e., control CVP 8-12 mmHg and give fluid when CVP < 8 mmHg.

Outcome analyses: Postoperative serum lactate and creatinine of both groups will be compared using unpaired Student-t test. Secondary outcomes will be compared using chi-square test.

ELIGIBILITY:
Inclusion Criteria:

1. 40-80 years old
2. Patient had aortic aneurysm both thoracic and abdominal types
3. Scheduled for elective EVAR procedures
4. New York Heart Association (NYHA) or American society of Anesthesiology (ASA) classification I-III
5. Body mass index (BMI) 18-24 kg/m2
6. Provided informed consent before surgery

Exclusion Criteria:

1. Scheduled for emergency or redo surgery
2. Received prior fluid therapy (>2,500 ml/day over the 48 h before the surgery)
3. Presence of congenital heart disease, cardiomyopathy, rheumatic heart disease, or significant arrhythmia or cardiopulmonary dysfunction, or significant renal or liver diseases
4. Preoperative use of vasoactive drugs (e.g. digoxin, nitroglycerine, nifedipine) for ≥3 months
5. Difficulty (or contraindication to) placing a central venous catheter
6. Inability to cooperate (e.g. mental disorder, disturbance of consciousness, mental retardation)
7. Presence of blood-borne infectious disease (e.g. syphilis, acquired immunodeficiency

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
lactate and creatinine level | at the end of surgery up to 48 hours
  serum lactate and creatinine level

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, Study Chair — Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramsingh DS, Sanghvi C, Gamboa J, Cannesson M, Applegate RL 2nd. Outcome impact of goal directed fluid therapy during high risk abdominal surgery in low to moderate risk patients: a randomized controlled trial. J Clin Monit Comput. 2013 Jun;27(3):249-57. doi: 10.1007/s10877-012-9422-5. Epub 2012 Dec 22. PMID 23264068
- [Result] Kothandan H, Haw Chieh GL, Khan SA, Karthekeyan RB, Sharad SS. Anesthetic considerations for endovascular abdominal aortic aneurysm repair. Ann Card Anaesth. 2016 Jan-Mar;19(1):132-41. doi: 10.4103/0971-9784.173029. PMID 26750684
- [Result] Brandstrup B. Fluid therapy for the surgical patient. Best Pract Res Clin Anaesthesiol. 2006 Jun;20(2):265-83. doi: 10.1016/j.bpa.2005.10.007. PMID 16850777